CLINICAL TRIAL: NCT05580783
Title: Iron Absorption and Variations of Iron Status Parameters, Hepcidin, Inflammatory Markers and Sex Hormones During the Menstrual Cycle
Brief Title: Iron Absorption and Variations of Iron Status, Hepcidin, Inflammation and Sex Hormones During the Menstrual Cycle
Acronym: MBL_Abs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Wageningen University and Research (Other); Sight and Life Foundation (Unknown); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Senior Scientist, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MBL_Abs; IZSTZ0_208432/1 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Iron-deficiency
Keywords: Anemia; Micronutrients; Iron; Trace elements; Menstruation; Hormones
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 54Fe (Experimental): Participants will receive 54Fe at two time points throughout their menstrual cycle.
  Interventions: Other: Test meal labelled with 54Fe
- Experimental 57Fe (Experimental): Participants will receive 57Fe at two time points throughout their menstrual cycle.
  Interventions: Other: Test meal labelled with 57Fe
- Experimental 58Fe (Experimental): Participants will receive 58Fe at two time points throughout their menstrual cycle.
  Interventions: Other: Test meal labelled with 58Fe

INTERVENTIONS:
Other: Test meal labelled with 54Fe — Each participant will receive 2 test meals containing 4mg each of isotopic tracer 54Fe
  Arms: Experimental 54Fe
Other: Test meal labelled with 57Fe — Each participant will receive 2 test meals containing 4mg each of isotopic tracer 57Fe
  Arms: Experimental 57Fe
Other: Test meal labelled with 58Fe — Each participant will receive 2 test meals containing 4mg each of isotopic tracer 58Fe
  Arms: Experimental 58Fe

SUMMARY:
Iron supplementation is the first line of treatment of iron deficiency in most women, but we do not know when the best time is to supplement in the context of the menstrual cycle. With this study, we aim to measure and compare iron status, hepcidin, inflammatory markers, hormones estrogen and progesterone and changes in iron absorption at various points throughout the menstrual cycle, with a long-term view to determine best time for iron supplementation in relation to the menstrual cycle.

DETAILED DESCRIPTION:
To date, very few studies have assessed iron absorption in relation to a woman's menstrual cycle. Although oral iron supplementation is considered the first line of treatment for iron deficiency in most women, there is no knowledge on the relationship between this intervention in the context of the menstrual cycle, and more specifically there is no knowledge on its potential implications for the most appropriate timing of iron supplementation. A better understanding of iron absorption during the menstrual cycle as well as kinetics of key parameters could allow the design of adapted and/or new interventions (e.g., timing of iron supplementation in relation to different phases of the menstrual cycle) to mitigate iron deficiency in menstruating women and can inform programs aimed at addressing iron deficiency

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-30 years old
* Weight <70 kg
* Normal body mass index (18.5 - 25kg/m2)
* Regular menstrual cycle (self-reported cycle length between 28 and 35 days in the past 6 months)
* Depleted iron stores (serum ferritin ≤ 30 µg/L)
* Signed informed consent
* Able to read and understand English

Exclusion Criteria:

* Use of hormonal contraceptives within a 3-month recall period
* Anemia (hemoglobin < 117 g/L)
* Any known major metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer, or cardiovascular diseases (according to the participants own statement)
* Women with severe menstrual cramps that would prevent them from attending study meetings during menstruation (judged by the women)
* Consumption of iron-containing supplements within 1 month prior to the start of study
* Known difficulties with blood sampling
* Pregnancy (serum human chorionic gonadotropin (hCG) < 5 mIU/mL)
* Current smoking (>1 cigarette per week over a 1-month recall period)
* Women who are planning to get pregnant within the study period, as this would affect iron metabolism and subsequent study measurements.
* Inability to follow the study protocol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption (%) | Day 2, 18, 22, 26 and 40
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the labelled test meals.

SECONDARY OUTCOMES:
Hemoglobin concentration (g/L) | Screening, day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28 and 40
  Haemoglobin will be measured to determine presence of anaemia
Serum ferritin (microg/L) | Screening, day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Iron status parameter
Serum transferrin receptor (mg/L) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Iron status parameter
Serum iron (microg/mL) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Iron status parameter
Serum hepcidin (nmol/L) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Hepcidin, a major regulator of iron absorption and influenced by inflammation, will be measured
Alpha-1-acid glycoprotein (g/L) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Chronic inflammation parameter
C-reactive protein (mg/L) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Acute inflammation parameter
Serum estradiol (pg/mL) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Hormonal parameter
Serum progesterone (ng/mL) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Hormonal parameter
Total iron binding capacity (microg/mL) | Day 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 28
  Total iron binding capacity will be measured to determine the presence of iron deficiency
Menstrual blood volume loss/cycle | Menstruation
  Semi-quantitative assessment to measure menstrual blood loss per cycle

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No